CLINICAL TRIAL: NCT03302481
Title: Prospective Physiopathology Study of the Links Between Mitochondrial Dynamics and Fatty Liver Disease During Obesity
Brief Title: Mitochondrial Metabolism and Hepatic Complications of Obesity
Acronym: DMSO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no ethic committee autorization
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC17_0055
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Obesity surgery; liver; mitochondria; steatosis
MeSH Terms: conditions — Obesity; Fatty Liver

STUDY DESIGN:
Intervention Model Description: patients with obesity surgery with a laparoscopic approach scheduled in the department of digestive surgery of the CHU de Nantes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): the biopsies will be performed under laparoscopy and taken in the lower part of the right hepatic lobe
  Interventions: Other: liver biopsy

INTERVENTIONS:
Other: liver biopsy — the biopsies will be performed under laparoscopy and taken in the lower part of the right hepatic lobe

SUMMARY:
The study aims to characterize mitochondrial metabolism in the liver of obesity surgery patients and to study its relationships with hepatic steatosis, inflammation, and fibrosis.

DETAILED DESCRIPTION:
The study aims to characterize mitochondrial metabolism in the liver of obesity surgery patients and to study its relationships with hepatic steatosis, inflammation, and fibrosis. The protocols involves a per-operative hepatic needle biopsy for mitochondria characterization and histological scoring of steatosis, inflammation, and fibrosis

ELIGIBILITY:
Inclusion Criteria:

* adult men and women
* affiliated to a social security
* candidate for laparoscopic obesity surgery

Exclusion Criteria:

* Excessive alcohol consumption:> 20 g / day (woman),> 30 g / day (male)
* Chronic viral hepatitis B or C
* Genetic hemochromatosis
* Taking the following drugs for at least 3 months up to 6 months before the scheduled date of obesity surgery: systemic corticosteroids, amiodarone, methotrexate
* Wilson's disease
* autoimmune hepatitis
* alpha 1-antitrypsin deficiency
* abetalipoproteinemia
* Contraindications to liver biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Association between nonalcoholic steato-hepatitis and mitochondria morphological markers | Until 6 month

CONTACTS AND LOCATIONS:
Overall Officials: David JACOBI, Dr, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: No